CLINICAL TRIAL: NCT00239083
Title: Phase IV Study of Efficacy and Safety of Enteric-Coated Mycophenolate Sodium (EC-MPS) in Combination With Cyclosporine Microemulsion (CsA-ME) in Kidney Transplant Patients
Brief Title: Efficacy and Safety of Enteric-Coated Mycophenolate Sodium (EC-MPS) in Renal Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080ATR01
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Kidney Transplantation
Keywords: MYFORMS, Kidney Transplantation, Enteric-Coated Mycophenolate Sodium (EC-MPS), Cyclosporine microemulsion (CsA-ME)

ARMS (1):
- EC-MPS (Experimental)
  Interventions: Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

SUMMARY:
The aim of MYFORMS is to assess efficacy and safety on clinical outcomes of EC-MPS in combination with Cyclosporine microemulsion (CsA-ME) in kidney transplant recipients.

ELIGIBILITY:
De Novo-Inclusion criteria

1. Males and females aged 6 years or over.
2. Recipients of cadaveric, living unrelated or living related kidney transplant, treated with CsA-Me, with or without corticosteroids, as primary immunosuppression.

Maintenance-Inclusion criteria

1. Males and females aged 6 years or over.
2. Recipients of first or secondary cadaveric, living related or unrelated donor kidney transplant.
3. Patients currently receiving CsA-ME with or without Mycophenolate mofetil (MMF) or azathioprine, with or without corticosteroids as part of their immunosuppressive regimen for at least 3 months prior to Screening.
4. Patients in a stable condition in terms of graft function (serum creatinine not above 2.3 mg/dL (=204 µmol/L) at screening and at baseline, or not increased by more than 20% at baseline compared to values obtained at screening), no change of immune suppressive regimen due to graft malfunction, and any known clinically significant physical and/or laboratory changes for at least 2 months prior to enrollment.

De Novo and Maintenance-Exclusion Criteria

1. Multi-organ recipients (e.g. kidney and pancreas) or previous transplant with any organ other than kidney.
2. Patients with any known hypersensitivity to MPA, EC-MPS or other components of the formulation (e.g. lactose).
3. Patients with thrombocytopenia (< 75,000/mm3), with an absolute neutrophil count of < 1,500/mm3, and/or leukocytopenia (< 2,500/mm3), and/or hemoglobin < 6 g/dL at Screening or Baseline.
4. Patients with a history of malignancy within the last five years, except excised squamous or basal cell carcinoma of the skin.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
patient and graft survival
acute rejection incidence
graft function
safety

SECONDARY OUTCOMES:
influence of demographic characteristics, transplant-related variables, medical conditions and post-transplantation complications on the main clinical outcomes, according to the immunosuppressive regimen used.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland

REFERENCES:
- [Result] Nart A, Sipahi S, Aykas A, Uslu A, Hoscoskun C, Toz H. Efficacy and safety of enteric-coated mycophenolate sodium in de novo and maintenance renal transplant patients. Transplant Proc. 2008 Jan-Feb;40(1):189-92. doi: 10.1016/j.transproceed.2007.11.066. PMID 18261583